CLINICAL TRIAL: NCT04789733
Title: Tight Perioperative Blood Pressure Management to Reduce Serious Cardiovascular, Renal, and Cognitive Complications: The GUARDIAN Pilot Trial
Brief Title: The GUARDIAN Pilot Trial
Acronym: GUARDIAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: The GUARDIAN pilot trial
Record Dates: First submitted 2021-01-14; First posted 2021-03-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: General Surgery
Keywords: Blood pressure; major adverse cardiac events; Delirium; Acute kidney injury
MeSH Terms: conditions — Cardiovascular Diseases; Delirium; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Parallel group randomized trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and assessors blinded to intraoperative management, postoperative antihypertensive management, and blood pressures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight pressure management (Experimental): Patients assigned to tight blood pressure control angiotensin converting enzyme inhibitors and angiotensin receptor blockers will not be given the morning of surgery. Other chronic antihypertensives will only be given as necessary to treat hypertension. Norepinephrine or phenylephrine infusion will be infused at a rate sufficient to maintain intraoperative MAP ≥ 85 mmHg.
  Resumption of chronic anti-hypertensive medications will be delayed until the third postoperative day unless deemed necessary to treat hypertension or for some other clear indication.
  The target for postoperative systolic arterial pressures ≥110 mmHg during the initial three postoperative days.
  Interventions: Other: Tight pressure management
- Routine pressure management (Other): ACEIs, ARBs, and/or calcium channel blockers can be given the morning of surgery if deemed appropriate by the attending anesthesiologist. Intraoperative blood pressure will be managed per clinical routine. As usual, chronic anti-hypertensive medications will be restarted shortly after surgery unless contraindicated by hypotension.
  Interventions: Other: Routine pressure management

INTERVENTIONS:
Other: Tight pressure management — Norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg, delayed resumption of chronic antihypertensive medications, and a target ward MAP ≥80 mmHg (tight pressure management)
  Arms: Tight pressure management
Other: Routine pressure management — Routine intraoperative blood pressure management and immediate restart of antihypertensive medications.
  Arms: Routine pressure management

SUMMARY:
The treatments will be: 1) norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg, delayed resumption of chronic antihypertensive medications, and a target ward MAP ≥80 mmHg (tight pressure management); or, 2) routine intraoperative blood pressure management and prompt resumption of chronic antihypertensive medications (routine pressure management).

DETAILED DESCRIPTION:
Consenting patients who take either angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), or calcium channel blockers will be asked not to take the medications on the morning of surgery, and instead bring them with them to the hospital. Qualifying patients will be randomized 1:1, with random-sized blocks.

Randomization will be implemented by clinicians in collaboration with research personnel. Arterial catheter transducers will be positioned at the level of the right atrium, and adjusted as necessary if patient position is changed.

The treatments will be: 1) norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg, delayed resumption of chronic antihypertensive medications, and a target ward MAP ≥80 mmHg (tight pressure management); or, 2) routine intraoperative blood pressure management and prompt resumption of chronic antihypertensive medications (routine pressure management).

Tight pressure management: In patients assigned to tight pressure management, angiotensin converting enzyme inhibitors and angiotensin receptor blockers will not be given the morning of surgery. Other chronic antihypertensives will only be given as necessary to treat hypertension. Clinicians will be encouraged to insert the required arterial catheter before anesthetic induction because much hypotension occurs shortly after anesthetic induction.

A norepinephrine or phenylephrine infusion (in the preferred local concentration) will be prepared, connected to an intravenous catheter, and activated at a low rate. Norepinephrine can be safely given through a central catheter or peripherally.

General anesthesia will be induced with propofol or etomidate which will be given in repeated small boluses or target-controlled infusion in an effort to keep mean arterial pressure ≥85 mmHg. Clinicians will be encouraged to use etomidate when rapid-sequence inductions are required. Simultaneously, the vasopressor infusion will be adjusted with the same goal. Anesthetic dose, fluid administration, and vasopressor administration will be adjusted with the goal of maintaining the individual designated baseline mean arterial pressure. Invasive or non-invasive advanced hemodynamic monitoring is not required, but should be used when practical. Clinicians should use available information to optimize vascular volume, afterload, and inotropy.

Resumption of chronic anti-hypertensive medications will be delayed until the third postoperative day unless deemed necessary to treat hypertension or for some other clear indication (e.g., preventing atrial fibrillation in a chronic beta-blocker user) because >90% of MINS occurs within 48 hours after surgery. When necessary to treat hypertension, chronic antihypertensive or new medications can be used per clinician preference. Clinicians will make what efforts they can to maintain postoperative mean arterial pressures ≥80 mmHg during the initial three postoperative days by maintaining adequate hydration, using inotropic and chronotropic drugs, and vasopressor as necessary. This protocol specifies the blood pressure target but leaves implementation to clinical judgement.

Routine pressure management: In patients assigned to routine pressure management, ACEIs, ARBs, and/or calcium channel blockers can be given the morning of surgery if deemed appropriate by the attending anesthesiologist. The arterial catheter will be inserted before or after induction of anesthesia per clinician preference. General anesthesia will be induced and maintained per routine. Blood pressure will not be deliberately reduced, but per routine clinicians will presumably not intervene until MAP is <65 mmHg. As usual, chronic anti-hypertensive medications will be restarted shortly after surgery unless contraindicated by hypotension.

In both groups, other aspects of anesthetic management will be at the discretion of the responsible anesthesiologist, including the types and volumes of various fluids. Volatile or intravenous anesthesia is permitted.

There will be no limitation on ancillary vasoactive, chronotropic, and inotropic drugs. Clinicians will be free to use advanced hemodynamic monitoring (e.g., pulse-wave analysis, esophageal Doppler, etc.). Blood products will be given per routine. Similarly, postoperative analgesic management will be per routine and clinician preference. Neuraxial and peripheral nerve blocks are permitted, but epidural catheters should not be activated until surgery is nearly finished.

Because patients must be fairly sick to qualify for GUARDIAN, some will go to directly from surgery to critical care units, or much less often, become unstable and require transfer from a routine ward to an ICU. In either case, every effort will be to maintain randomized treatments and blood pressure targets.

In all cases, good judgement will predominate. Clinicians should always act in their patients' best interests, irrespective of the GUARDIAN protocol

ELIGIBILITY:
Inclusion Criteria:

* ≥45 years old
* Scheduled for major noncardiac surgery expected to last at least 2 hours;
* Having general endotracheal, neuraxial anesthesia, or the combination;
* Expected to require at least overnight hospitalization;
* Are designated ASA physical status 2-4 (ranging from mild systemic disease through severe systemic disease that is a constant threat to life);
* Chronically taking at least one anti-hypertensive medication;
* Expected to have direct blood pressure monitoring with an arterial catheter;
* Cared for by clinicians willing to follow the GUARDIAN protocol;
* Subject to at least one of the following risk factors:
* History of peripheral arterial surgery;
* History of coronary artery disease;
* History of stroke or transient ischemic attack;
* Serum creatinine >175 µmol/L (>2.0 mg/dl);
* Diabetes requiring medication;
* Current smoking or 15 pack-year history of smoking tobacco;
* Scheduled for major vascular surgery;
* Body mass index ≥35 kg/m2;
* Preoperative high-sensitivity troponin T >14 ng/L or troponin I equivalent;
* B-type natriuretic protein (BNP) >80 ng/L or N-terminal B-type natriuretic protein (NT-ProBNP) >100 ng/L

Exclusion Criteria:

* Are scheduled for carotid artery surgery;
* Are scheduled for intracranial surgery;
* Are scheduled for partial or complete nephrectomy;
* Are scheduled for pheochromocytoma surgery;
* Are scheduled for liver transplantation;
* Require preoperative intravenous vasoactive medications;
* Have a condition that precludes routine or tight blood pressure management such as surgeon request for relative hypotension;
* Require beach-chair positioning;
* Have end-stage renal disease requiring dialysis or estimated glomerular filtration rate (eGFR) <30 ml/min;
* Have a documented history of dementia;
* Have language, vision, or hearing impairments that may compromise cognitive assessments;
* Have contraindications to norepinephrine or phenylephrine per clinician judgement;
* Have previously participated in this trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood pressure management | Intraoperative
  The fraction of time when intraoperative MAP is <65 mmHg and ≥85 mmHg during surgery.
Postoperative blood pressure management | First 3 postoperative days
  Time to restarting routine antihypertensive medications.

SECONDARY OUTCOMES:
Intraoperative pressure | Intraoperative
  Time-weighted mean-arterial pressure
Postoperative pressure | Initial 3 postoperative days
  Time-weighted systolic pressure

OTHER OUTCOMES:
Perfusion-related complications | 30 days
  A composite of serious perfusion-related complications: myocardial injury, stroke, non-fatal cardiac arrest, Stage 2-3 acute kidney injury, deep or organ-space infection, sepsis, and death.
Delirium | Initial 4 postoperative days
  Postoperative delirium assessed with 3D CAM ICU twice daily.

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Union Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Li K, Hu Z, Li W, Shah K, Sessler D. Tight perioperative blood pressure management to reduce complications: a randomised feasibility trial. BMJ Open. 2023 Nov 17;13(11):e071328. doi: 10.1136/bmjopen-2022-071328. PMID 37977865